CLINICAL TRIAL: NCT03851718
Title: Effect of Acupuncture on Hypogalactia (Decreased Milk Supply): A Pilot Study
Brief Title: Effect of Acupuncture on Hypogalactia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI leaves the study institution.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L18-195
Record Dates: First submitted 2019-02-14; First posted 2019-02-22 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Hypogalactia
Keywords: Acupuncture; Hypogalactia; Power Pumping; Brest Milk Production
MeSH Terms: conditions — Lactation Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Acupuncture Procedure (Experimental): Acupuncture is a type of Traditional Chinese Medicine (TCM) therapeutic approaches involving the insertion and manipulation of fine needles in specific points. Mothers in acupuncture group will be given three standardized sessions of acupuncture within 5 weekdays, preferably on 3 consecutive days.
  Interventions: Device: Acupuncture Procedure
- Power pumping (Active Comparator): Power pumping is a pumping strategy that mimics normal infant cluster feedings by repeatedly emptying mother's breast very frequently in an effort to increase breast milk supply. As there is no standardized protocol of power pumping, one of the most popular recommendations will be adapted as the study power pumping instruction. It suggests the mom to set at least one hour and two hours preferably for the power pumping at least three days within a 5 weekday period, preferably on 3 consecutive days.
  Interventions: Behavioral: Power pumping

INTERVENTIONS:
Device: Acupuncture Procedure — Each session will run about 30~40 minutes at the Family Medicine Clinic and performed by a licensed acupuncturist. The expense of all three sessions will be reimbursed by the project, not billed to the participant. The following points CV17, ST18 (bilateral), ST36 (bilateral), SI1(bilateral) and LR3(bilateral) , adopted from TCM classic text and previous studies done in China, will be used for all three sessions .
  Arms: Acupuncture Procedure
Behavioral: Power pumping — It suggests the mom to set at least one hour and two hours preferably for the power pumping at least three days within a 5 weekday period, preferably on 3 consecutive days. During this one hour, the moms will be advised to pump for 20 minutes, rest for 10 minutes, pump for 10 minutes, then rest for 10 minutes and pump for 10 minutes. Alternatively they can also opt to pump and rest for every 10 minutes during the hour.
  Arms: Power pumping

SUMMARY:
The specific aims are (1) to assess the feasibility of a RCT studying acupuncture's impact on breast milk production, and (2) to compare the difference of milk production between acupuncture and power pumping. The study approach will be a two-site prospective, non-blinded, two-arm randomized clinical trial conducted in Lubbock and Amarillo as a collaborative effort between researchers and clinicians in the departments of Family Medicine, Pediatrics and Ob/Gyn. An estimated 60 eligible mothers will be recruited and enrolled in the study from both sites. The participants will be randomized 1:1 into either the intervention group or the comparison group. The intervention group will receive three standardized acupuncture sessions, based on previous studies done in China and investigators' practice protocol, in 5 days and the comparison group will perform power pumping in 5 days per provided manual and guidance. The primary outcome is changes of breast milk production and it will be measured by weighing the grams/volume of milk expressed with an electric breast pump over time. The secondary outcome is changes of plasma prolactin and it will be measured by immunoassay. Data will be collected at baseline, right after interventions and two week after interventions to compare the difference of the outcomes. The findings of this study will provide insight to establish a RCT protocol to assess acupuncture's impact on hypogalactia. It may also help establish evidence of acupuncture use for hypogalactia.

DETAILED DESCRIPTION:
As important and beneficial as breastfeeding is to infants and mothers, physicians often feel lack resources to support breast milk production. Reduced breast milk production (called hypogalactia) is the most frequent cause of breastfeeding failure, but no evidenced-based standard care in conventional medicine is established to help mothers face the challenge. The most frequently used natural galactogogues products including galega and silymarin are not FDA approved. Lactation education on general breastfeeding and lactation management may help mothers who are experiencing reduced milk supply. Complementary and alternative medicine (CAM) including acupuncture has been used to address hypogalactia. However, there remains an overall lack of evidence regarding the effectiveness, safety, and acceptability of many CAM therapies including acupuncture for hypogalactia. Although several clinical observational studies showed that acupuncture was related to the increased prolactin level and mother's breast milk production, there are several gaps in those studies. First, most studies were done in China and are mainly observational, hence are subject to various biases and do not establish a causal relationship. Secondly, most of the studies only reported success rates without reporting changes of milk volume or biomarkers. To truly assess the effect of acupuncture on breast milk production and relevant hormone changes, a randomized clinical trial (RCT) with better measurements is warranted.

The feasibility of an acupuncture protocol for hypogalactia is supported by the acupuncture practice in the Family medicine clinic. The goal of this study is to establish the feasibility of a RCT to compare the difference of breast milk production between acupuncture and power pumping, a popular lactation practice recommended to mothers who experience hypogalactia, using established measurement of breast milk production. Both acupuncture and power pumping stimulate the breasts which may lead to the increased secretion of prolactin hence increase milk production. Previous study findings and investigators' clinical experiences indicate that a short period of acupuncture treatment may increase milk production for several weeks. It is hypothesized that acupuncture will have equal or a greater impact on milk production and last longer than power pumping. The study special aims are:

1. To assess the feasibility of a RCT studying acupuncture's impact on breast milk production. A two-arm RCT will be conducted at one site. Recruitment, enrollment, intervention and compliance, safety and adverse events will be documented and evaluated to assess this trial design is appropriate for further testing. Study feasibility is defined as the successful recruitment and retention of study participants, adherence to the intervention, identification of barriers to the intervention, and the rigorous collection of outcome data.
2. To compare the effect difference of breast milk production between acupuncture and power pumping. The primary outcome the changes of breast milk production will be measured by weighing the grams/volume of milk expressed with an electric breast pump. The secondary outcome the changes of plasma prolactin will be measured by immunoassay. Data will be collected at baseline, right after interventions and two week after interventions.

Based on investigators' search in PubMed to present, no RCT studies have been done in the U.S. assessing acupuncture and hypogalactia. This study may be the first to provide insights on the feasibility. Moreover, based on investigators's clinical observations and reports from studies done in China, this study to yield positive findings to help establish evidence of acupuncture use for hypogalactia. The preliminary data may also help us apply for grants from the National Center for Complementary and Integrative Health (NCCIH) or NIH Office of Research on Women's Health. More importantly, the evidence will help clinician and mothers make informed decisions in terms of choosing the right approach to increase breast milk production.

ELIGIBILITY:
Inclusion Criteria:

1. Primipara or Multipara woman who had normal pregnancy (gestation ≥ 37 weeks gestation) and gave birth vaginally or by Caesarean section to a single child without complications and who are 2 weeks to 6 months postpartum.
2. Estimated milk production of < 450 g/24 hours (or 450ml/24hours)-by self-report
3. A current body mass index (BMI) equal or above 18 kg/m2 and below 35 kg/ m2
4. Non-smoker. Subjects who have stopped smoking for >6 months prior to study start may be included.
5. Must be fluent in English conversation, reading and writing.

Exclusion Criteria:

1. Presence or a history of clinically significant diseases of the renal, hepatic, gastrointestinal, cardiovascular, musculoskeletal systems or presence or history of clinically significant psychiatric, immunological, endocrine or metabolic diseases including gestational or pregestational diabetes, and Polycystic Ovarian syndrome.
2. History of breast cancer, breast surgery, or clinically significant abnormalities of the breasts that may affect the milk production and/or flow.
3. Use of typical and atypical antipsychotics, drugs/supplements, and/or other approaches that may increase milk production or prolactin levels in patients.
4. Consumes alcohol during breastfeeding.
5. Current case of infectious mastitis and/or Reynaud's disease of the breast.
6. History within the last two years or current abuse of alcohol or drugs.
7. Current non-smokers with a history of long-term, heavy smoking (>10 pack-years).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
changes of breast milk production volume from based line to within 48 hours after the last intervention session. | Measurements will be done during the study at baseline and right after (i.e. within 48 hours) after last acupuncture session or power pumping secession.
  Breast Milk Production will be measured by weighing the grams/volume of milk expressed with an electric breast pump (e.g. Spectra Baby USA) at four sequential hourly intervals including zero time.
changes of breast milk production volume from based line to at 2 weeks after the last intervention session. | Measurements will be done during the study at baseline and 2 weeks after last acupuncture session or power pumping secession.
  Breast Milk Production will be measured by weighing the grams/volume of milk expressed

SECONDARY OUTCOMES:
changes of prolactin level from based line from based line to within 48 hours after the last intervention session. | Measurements will be done during the study at baseline and right after (i.e. within 48 hours) after last acupuncture session or power pumping secession.
  the participants will have 7 ml of blood drawn by venipuncture utilizing a serum separator tube. A blood collection log and labels will be created. The sample will be taken to the laboratory, allowed to clot and then centrifuged at 2500-3200 rpm for 5-6 minutes to separate the serum from the cells. Samples will be analyzed for prolactin using a Beckman Coulter Access 2 Immunoassay Analyzer and an FDA approved in vitro diagnostic Prolactin assay kit according to clinical standards.
changes of prolactin level from based line to 2 weeks after the last intervention session. | Measurements will be done during the study at baseline and 2 weeks after last acupuncture session or power pumping secession.
  the participants will have 7 ml of blood drawn by venipuncture utilizing a serum separator tube. A blood collection log and labels will be created. The sample will be taken to the laboratory, allowed to clot and then centrifuged at 2500-3200 rpm for 5-6 minutes to separate the serum from the cells. Samples will be analyzed for prolactin using a Beckman Coulter Access 2 Immunoassay Analyzer and an FDA approved in vitro diagnostic Prolactin assay kit according to clinical standards.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is not a plan to make individual participant data (IPD) available to other researchers at this time.